CLINICAL TRIAL: NCT07379671
Title: The Effect of the Mamelon Effect on Upper Incisors on the Perception of Smile Esthetics
Brief Title: The Effect of the Mamelon Effect on the Perception of Smile Esthetics
Acronym: MamelonEffect
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: BK_MarmaraU
Record Dates: First submitted 2026-01-13; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Restorative Experiences; Esthetic Restorations; Perception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group/Cohort 1: Laypeople: Laypersons with no formal dental education who participated in the online survey to evaluate digitally modified smile images. Participants assessed the esthetic attractiveness of full-face and close-up smile photographs using a visual analog scale (VAS).
  Interventions: Other: Online Survey
- Group/Cohort 2: Dentists: General dentists who participated in the online survey and evaluated digitally modified smile images. Participants assessed the esthetic perception of different incisal mamelon configurations using a visual analog scale (VAS).
  Interventions: Other: Online Survey
- Group/Cohort 3: Dental Specialists: Dental specialists in Restorative Dentistry and Prosthodontics who participated in the online survey. Participants evaluated digitally modified smile images with varying mamelon characteristics using a visual analog scale (VAS).
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — An anonymous web-based survey was used to assess the perception of smile esthetics. Participants evaluated a total of 18 images (including original and digitally modified full-face and close-up images) using a visual analog scale ranging from 0 (extremely unattractive) to 100 (extremely attractive).

SUMMARY:
This study aimed to evaluate the role of the mamelon effect on the perception of smile esthetics. A single portrait image was digitally modified by using the Photoshop CC (Adobe, USA) software program to create the mamelon effects at the incisal edge of maxillary incisors. Length (cervico-incisal) and value (level of gray color) were the variables in the modified images. There were two length (1mm and 3mm) and two value (low value, LV and high value, HV) modifications performed for the central incisors (2 teeth) and for the central and lateral incisors together (4 teeth). Eight full-face and 8 close-up images were created by cropping the modified images. In total 18 images (including the original ones) were evaluated by the participants. 135 participants (45 dentists, 45 specialists, and 45 laypeople) contributed to an online survey to evaluate the digitally modified images by using a visual analog scale ranging from 0 - 100, according to their level of attractiveness. The data were analyzed using Bonferroni Pairwise Comparisons. The results were presented as average±standard deviation. The deemed significance was set at <.050.

DETAILED DESCRIPTION:
This observational, cross-sectional study was designed to investigate the effect of incisal mamelon characteristics on the perception of smile esthetics using digitally modified facial images. The study protocol was approved by the Marmara University Faculty of Medicine Ethics Committee and was conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines. Written informed consent was obtained from the volunteer whose facial photographs were used, as well as from all survey participants.

Study Design and Image Preparation A single volunteer meeting the inclusion criteria (aged 18-65 years; clinically healthy maxillary anterior teeth; proportional tooth dimensions; no restorations, orthodontic anomalies, or pronounced mamelon appearance) was selected. Extraoral smile photographs were captured using a digital single-lens reflex (DSLR) camera under standardized lighting conditions. Both full-face smile and close-up smile images were obtained to reflect different viewing distances relevant to daily social interactions and clinical evaluations.

The original digital image was transferred to a computer environment and edited using image-processing software (Adobe Photoshop CC, Adobe Systems, USA). Digital modifications were limited to the maxillary incisors (central and lateral teeth) while preserving facial symmetry, dental midline, gingival contours, and surrounding oral tissues.

Two main variables were manipulated:

Mamelon length (cervico-incisal extension): 1 mm and 3 mm Mamelon value (brightness level): low value (LV) and high value (HV) Mamelon effects were applied either to the maxillary central incisors alone (2 teeth) or to both central and lateral incisors simultaneously (4 teeth). Using these parameters, digitally modified images were created to simulate different mamelon configurations while maintaining natural tooth anatomy and proportions.

Study Groups and Image Sets

A total of 16 modified images were generated from the original photograph, consisting of:

8 full-face smile images 8 close-up smile images Together with the original unmodified full-face and close-up images, a total of 18 images were included in the evaluation set. All images were randomized prior to assessment to minimize ordering and learning effects.

Participants and Survey Procedure

A total of 135 participants were recruited and equally distributed into three observer groups:

Dentists (n = 45) Dental specialists (restorative dentistry and prosthodontics) (n = 45) Laypersons with no dental education (n = 45) Participants completed an anonymous online survey. Demographic information including age, gender, and professional background was recorded. Each participant evaluated all 18 images using a visual analog scale (VAS) ranging from 0 to 100, where higher scores indicated greater perceived smile attractiveness.

Outcome Measures

The primary outcome measure was the perceived smile esthetic score assigned to each image. Secondary analyses examined the influence of:

Image type (full-face vs. close-up) Mamelon length Mamelon value Number of teeth involved (2 vs. 4 incisors) Observer group (dentists, specialists, laypersons) Gender of the observers Statistical Analysis Statistical analysis was performed using appropriate statistical software. Descriptive statistics were calculated as mean ± standard deviation. Pairwise comparisons between groups and image conditions were conducted using Bonferroni-adjusted post hoc tests. The level of statistical significance was set at p < 0.05.

Ethical Considerations All photographic materials were obtained following written informed consent, including explicit permission for digital modification and scientific use of the images. Survey participation was voluntary and anonymous. No financial compensation was provided. The study involved no clinical intervention, and no risks beyond routine survey participation were anticipated.

Clinical Relevance By evaluating the esthetic impact of digitally simulated mamelon variations under different viewing conditions and observer profiles, this study aims to provide clinically relevant guidance for anterior restorative treatment planning. Understanding how mamelon characteristics influence esthetic perception may assist clinicians in making more patient-centered decisions regarding incisal anatomy in esthetic restorations

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ability to understand the study information and provide informed consent
* Participation on a voluntary basis
* Completion of the online survey only once
* Belonging to one of the following observer groups:
* Laypersons with no dental education
* Licensed dentists
* Dental specialists in Restorative Dentistry or Prosthodontics

Exclusion Criteria:

* Age <18 years
* Inability to understand the study information or provide informed consent
* Incomplete survey response
* Multiple survey submissions by the same participant
* Participation outside the predefined observer groups
* People with mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 135 adult participants were included in the study. The study population comprised equal numbers of laypersons, licensed dentists, and dental specialists in Restorative Dentistry or Prosthodontics (n = 45 per group).
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Perception of smile esthetics with different incisal mamelon configurations | Approximately 10-15 minutes
  Participants were asked to evaluate the esthetic attractiveness of digitally modified smile images presenting different incisal mamelon configurations. Evaluations were performed using a visual analog scale (VAS) ranging from 0 (extremely unattractive) to 100 (extremely attractive). The influence of mamelon length (1 mm vs 3 mm), mamelon value (low vs high), and the number of teeth involved (2 incisors vs 4 incisors) on esthetic perception was assessed.

SECONDARY OUTCOMES:
Effect of image type on esthetic perception | Approximately 10-15 minutes
  The esthetic perception scores of full-face smile images were compared with close-up smile images to evaluate the effect of viewing distance on the perception of incisal mamelon characteristics. Evaluations were performed using a visual analog scale (VAS) ranging from 0 to 100.
Effect of observer group on esthetic perception | Approximately 10-15 minutes
  Differences in esthetic perception scores among laypersons, dentists, and dental specialists were analyzed to assess the influence of professional background on the evaluation of incisal mamelon characteristics. All images were rated using a Visual analog scale (minimum 0, maximum 100). As the score increases, the aesthetic perception value increases.
Effect of observer gender on esthetic perception | Approximately 10-15 minutes
  Esthetic perception scores were compared according to the gender of the observers to evaluate potential differences in the perception of digitally simulated incisal mamelon effects. Ratings were obtained using a visual analog scale (minimum 0, maximum 100). As the score increases, the aesthetic perception value increases.
Interaction between mamelon length and value on esthetic perception | Approximately 10-15 minutes
  The combined effect of mamelon length (1 mm vs 3 mm) and mamelon value (low vs high) on smile esthetic perception was evaluated based on Visual Analog Scale scores obtained from all participant groups. Visual analog scale (minimum 0, maximum 100). As the score increases, the aesthetic perception value increases.

CONTACTS AND LOCATIONS:
Overall Officials: Bora Korkut, Assoc. Prof. Dr., Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.
Supporting Information: Study Protocol